CLINICAL TRIAL: NCT04841785
Title: The RECOVAC LESS CoV-2 Study - Long Term Efficacy and Safety of SARS-CoV-2 Vaccination in Patients in Patients With Chronic Kidney Disease Stage G4-G5, on Dialysis or After Kidney Transplantation
Brief Title: RECOVAC - Long Term Efficacy and Safety of COVID-19 (SARS-CoV-2) Vaccination in Kidney Disease Patients
Acronym: LESS CoV-2
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, J.S.F. Sanders, Study coordinator, University Medical Center Groningen
Other Study IDs: NL76839.042.21
Record Dates: First submitted 2021-03-22; First posted 2021-04-12 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Covid19; SARS-CoV Infection; Chronic Kidney Diseases
Keywords: Kidney transplant recipients; Dialysis; Chronic kidney disease stage 4-5; SARS-CoV-2 vaccination; COVID-19 vaccination; Antibody based immune response
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (in total maximum 1 mL) with a mailer-based finger-prick will be drawn
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CKD4/5: Patients with chronic kidney disease stage G4-G5 without dialysis or with a kidney transplant
  Interventions: Diagnostic Test: mailer-based finger-prick
- Dialysis: Patients on hemodialysis and peritoneal dialysis
  Interventions: Diagnostic Test: mailer-based finger-prick
- Kidney transplant: Patients with a kidney transplant at least 6 weeks after transplantation
  Interventions: Diagnostic Test: mailer-based finger-prick

INTERVENTIONS:
Diagnostic Test: mailer-based finger-prick — All participants in the antibody measurement study will be sent a mailer-based finger-prick set. The sets will be sent to the home address of the patient, including a return envelope. After collecting and returning the samples SARS-CoV-2 antibodies will be analysed quantitatively at the laboratory.
  Other Names: blood withdrawel

SUMMARY:
Rationale: COVID-19 is associated with severely increased morbidity and mortality in patients with chronic kidney disease stage G4-G5 and patients on dialysis or after kidney transplantation. Therefore, effective SARS-CoV-2 vaccination would be of great clinical importance in these patients. However, SARS-CoV-2 vaccination studies have excluded these patients so-far. Literature data indicate that vaccination may be less effective in these patient groups.

Objective: To assess the efficacy and safety of SARS-CoV-2 vaccination in patients with chronic kidney disease stage G4-G5, patients on dialysis or after kidney transplantation during two years follow-up after vaccination.

Study design: prospective single center observational cohort study.

Study population:

* all Dutch patients on dialysis with data registered in the Dutch Dialysis registry (RENINE)
* all Dutch patients after kidney transplantation with data registered in the Dutch national kidney transplant registry (NOTR).
* All Dutch patients with chronic kidney disease stage G4-G5 registered in the Santeon hospitals.

Intervention: After SARS-CoV-2 vaccination according to standard of care, blood will be drawn for antibody response measurements at day 28 and month 6 after 2nd vaccination at by mailer-based finger-prick in 3400 hemodialysis patients, 600 peritoneal dialysis patients, 4000 patients after kidney transplantation and 4000 patients with chronic kidney disease stage G4-G5. Patients who will undergo a 3rd SARS-CoV-2 vaccination via the national vaccination program for immunocompromised patients will be asked to carry out the mailer-based finger-prick 28 days after the 3rd SARS-CoV-2 vaccination, instead of the antibody measurement 6 months after the 2nd SARS-CoV-2 vaccination.

Main study parameters/endpoints:

The primary endpoint is efficacy of SARS-CoV-2 vaccination determined as:

- the incidence of COVID-19 after vaccination.

Secondary endpoints are

* mortality
* adverse events of specific interest according to (inter)national authorities in collaboration with LAREB
* presence of HLA-antibodies in dialysis patients on the waiting list for a first kidney transplantation
* acute rejection and graft failure in patients after kidney transplantation In a subset of patients additional secondary endpoints will be assessed
* the antibody based immune response at 28 days after completion of SARS-CoV-2 vaccination.
* the durability of antibody based immune response at 6 months compared to at 28 days after having received two subsequent SARS-CoV-2 vaccinations, in patients that have not received a 3rd SARS-CoV-2 vaccine.
* the antibody based immune response at 28 days after having received the 3rd SARS-CoV-2 vaccination.

The incidence of these endpoints will be compared, if applicable, to those:

* in the general population who are vaccinated
* in patients on dialysis or after kidney transplant who are not vaccinated Within these patient groups endpoints will be compared between recipients of different vaccines.

DETAILED DESCRIPTION:
1. OBJECTIVES

   Primary objective:

   To assess the efficacy of SARS-CoV-2 vaccination by the incidence of COVID-19 in patients with chronic kidney disease stage G4-G5, on dialysis and patients after kidney transplantation who received SARS-CoV-2 vaccination

   Secondary Objectives:

   - To assess the safety of vaccination

   In a subgroup of participants:
   * To assess the level of antibody response at 28 days and 6 months after SARS-CoV-2 vaccination
   * To assess durability of the antibody response at 6 months after having received two subsequent SARS-CoV-2 vaccinations, in a subset of patients that have not received a 3rd SARS-CoV-2 vaccine
   * the antibody based immune response at 28 days after having received the 3rd SARS-CoV-2 vaccination.

   Exploratory Objectives:
   * The vaccination coverage rate
   * The severity of COVID-19 in case of infection
   * The influence of vaccination on health-related quality of life by patient reported outcome measures (PROMs) in patients on dialysis.
   * The SARS-CoV-2 genotype in patients with COVID-19

   In a subgroup of participants:
   * To assess the level of antibody response after vaccination between patients with COVID-19 and without COVID-19 at:

     * 28 days after the 2nd SARS-CoV-2 vaccination
     * 28 days after the 3rd SARS-CoV-2 vaccination
     * 6 months after the 2nd SARS-CoV-2 vaccination in patients who have not received a 3rd vaccine.
   * To assess change in behaviour towards measures against COVID-19 before and after vaccination

   If data are available and applicable, outcomes in vaccinated patients on dialysis or after kidney transplantation will be compared:
   * with outcomes in the general population
   * with outcomes in patients with severely impaired kidney function (CKD stages G4/5), on dialysis or with a kidney transplant who are not vaccinated.
   * according to the type of vaccination they received
2. STUDY DESIGN

   This is a prospective observational registry-based cohort study to evaluate the long-term efficacy and safety after SARS-CoV-2 vaccination on clinically important outcomes in patients with chronic kidney disease stage G4-G5, on dialysis or after kidney transplantation.

   All participants will receive vaccination against COVID-19 via the national vaccination program and according to the manufacturer's instructions. To assess the immune response after vaccination, blood samples will be collected at 28 days after the 2nd SARS-CoV-2 vaccination, 28 days after the 3rd SARS-CoV-2 vaccination, and 6 months after the 2nd SARS-CoV-2 vaccination in patients who have not received a 3rd vaccination. In total a maximum of 1 ml blood will be drawn.

   Data of the following cohorts will be analyzed in this study.
   * Patiens with chronic kidney disease stage G4-G5, data to be derived from the Santeon hospitals.
   * Patients on hemodialysis and peritoneal dialysis, data to be derived from the existing national registry RENINE
   * Kidney transplant recipients, data to be derived from the existing national registry NOTR
   * Patients on dialysis or after kidney transplantation with COVID-19 disease, data to be derived from the ERACODA database.
3. METHODS

Main study parameter/endpoint:

The primary endpoints is the incidence of COVID-19 in a two years period after SARS-CoV-2 vaccination in patients with chronic kidney disease stage G4-G5, on dialysis or after kidney transplantation.

Secondary study parameters/endpoints:

Safety in all patients:

* Incidence of mortality
* Incidence of adverse events of specific interest as defined by (inter)national authorities in collaboration with LAREB
* Incidence of a combined endpoint of acute rejection or graft failure in patients after kidney transplantation
* Incidence of HLA antibodies defined as calculated Panel Reactivity Antibodies (cPRA) > 5% in patients on the waiting list for their first kidney transplantation

Efficacy in a subgroup of patients:

* The antibody response against the SARS-CoV-2 Receptor Binding Domain at 28 days after the final SARS-CoV-2 vaccination.
* The antibody response against the SARS-CoV-2 Receptor Binding Domain at 28 days after the 3rd SARS-CoV-2 vaccination.
* The durability of antibody based immune response against SARS-CoV-2 Receptor Binding Domain at 6 months compared to 28 days after completion of SARS-CoV-2 vaccination in patients who did not receive a 3rd SARS-CoV-2 vaccination.

Exploratory study parameters:

* Vaccination coverage rates
* Disease severity in patients who develop COVID-19, assessed as
* Hospitalization
* ICU admission
* Mechanical ventilation
* Mortality
* The influence of vaccination on health-related quality of life by patient reported outcome measures (PROMs) in dialysis patients
* SARS-CoV-2 genotype in patients with COVID-19

In a subgroup of participants:

* To assess the level of SARS-CoV-2 Receptor Binding Domain antibody response after vaccination between patients with COVID-19 and without COVID-19 at:

  * 28 days after the 2nd SARS-CoV-2 vaccination
  * 28 days after the 3rd SARS-CoV-2 vaccination
  * 6 months after the 2nd SARS-CoV-2 vaccination in patients who have not received a 3rd vaccine.
* To assess change in behaviour towards measures against COVID-19 before and after vaccination

These data collected after SARS-CoV-2 vaccination in patients with chronic kidney disease stage G4-G5, on dialysis and after a kidney transplantation will (if applicable data are available) be compared:

* to those obtained in the general population
* to those obtained in patients with chronic kidney disease stage G4-G5, on dialysis or with a kidney transplant who are not vaccinated
* according to the type of vaccination received These comparisons will allow us to analyze whether SARS-CoV-2 vaccination offers efficacy to prevent COVID-19 and sufficient safety in patients with chronic kidney disease stage G4-G5, dialysis and kidney transplant patients when compared to non-vaccinated patients with chronic kidney disease stage G4-G5, dialysis and kidney transplant patients, whether the efficacy is similar as in the general population, and whether there are differences in the risk-benefit ratio between the various vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for COVID-19 vaccination as described by the instructions of the manufacturer.
2. Age of 18 years or older
3. Capable of understanding the purpose and risks of the study, fully informed and given written informed consent (signed informed consent form has been obtained)
4. Either

   * eGFR < 30 ml/min/1.73m2 but not on dialysis or with a kidney transplant
   * Hemodialysis, or peritoneal dialysis
   * Kidney Transplant recipient at least 6 weeks after transplantation

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g. anaphylaxis) to any component of the study intervention(s).
* Patients who opted out for research in the Santeon, RENINE and NOTR registries.
* Patients who participate in the RECOVAC-IR study.
* Of note, patients will be eligible whether or not they have a history of COVID-19. Analyses will be performed in the overall population, but also shown separately for those without and with a history of COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with chronic kidney disease stage G4-G5 from the Santeon registry
  * Patients on hemodialysis and peritoneal dialysis who gave informed consent for participating in the national registry RENINEKidney transplant recipients who gave informed consent for participating in the national registry NOTR
Sampling Method: Probability Sample
Enrollment: 4868 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
The incidence of COVID-19 | two years after SARS-CoV-2 vaccination
  After SARS-CoV-2 vaccination in patients with chronic kidney disease stage G4-G5, on dialysis or after kidney transplantation.

SECONDARY OUTCOMES:
Incidence of mortality | two years after SARS-CoV-2 vaccination
  Incidence of mortality in patients with chronic kidney disease stage G4-G5, on dialysis or after kidney transplantation.
Incidence of adverse events | two years after SARS-CoV-2 vaccination
  Incidence of adverse events of specific interest as defined by (inter)national authorities in collaboration with LAREB
Incidence of acute rejection or graft failure in kidney transplant recipients | two years after SARS-CoV-2 vaccination
  Incidence of a combined endpoint of acute rejection or graft failure in patients after kidney transplantation
Incidence of HLA antibodies measured in blood | two years after SARS-CoV-2 vaccination
  Incidence of HLA antibodies defined as calculated Panel Reactivity Antibodies (cPRA) > 5% in patients on the waiting list for their first kidney transplantation
The antibody level against the SARS-CoV-2 Receptor Binding Domain measured in blood | 28 days after second SARS-CoV-2 vaccination.
  The antibody response against the SARS-CoV-2 Receptor Binding Domain
The antibody level against SARS-CoV-2 Receptor Binding Domain measured in blood | 6 months after second SARS-CoV-2 vaccination
  The antibody based immune response against SARS-CoV-2 Receptor Binding Domain at 6 months compared to 28 days after completion of SARS-CoV-2 vaccination in patients without a third vaccination.
The antibody level against SARS-CoV-2 Receptor Binding Domain measured in blood | 28 days after third SARS-CoV-2 vaccination
  The antibody based immune response against SARS-CoV-2 Receptor Binding Domain at 28 days after a third vaccination

OTHER OUTCOMES:
Vaccination coverage rate | two years
  Percentage of patients vaccinated
SARS-CoV-2 genotype | two years
  In patients with active COVID-19 infection
Level of SARS-CoV-2 Receptor Binding Domain antibody in patients with and without COVID-19 | two years
  level of SARS-CoV-2 Receptor Binding Domain antibody response at 28 days and 6 months after the second SARS-CoV-2 vaccination (in patients who did not receive a third vaccination) or 28 days after the third SARS-CoV-2 vaccination between patients who develop COVID-19 and who do not develop COVID-19 after vaccination
Disease severity of COVID-19 in case of infection assessed by ICU admission | two years
  Number of ICU admissions with COVID-19 after vaccination
Disease severity of COVID-19 in case of infection assessed by mechanical ventilation | two years
  Number of cases with mechanical ventilation because of COVID-19 after vaccination
Disease severity of COVID-19 in case of infection assessed by mortality | two years
  Number of deaths due to COVID-19 after vaccination
Disease severity of COVID-19 in case of infection assessed by hospitalization | two years
  Number of hospital admissions with COVID-19 infection after vaccination
Influence of vaccination on health related quality of life - SF-12 | two years
  Measured by Patient Reported Outcome Measures (PROMs). This is a questionnaire consisting of two parts. The first part includes the 12 items Short Form (SF-12) health survey to monitor physical and mental quality of life (with a score on 8 categories ranging from 0-100; with a higher score defined as a higher quality of life). Scores before and after vaccination will be compared.
Influence of vaccination on health related quality of life - DSI | two years
  Measured by Patient Reported Outcome Measures (PROMs). This is a questionnaire consisting of two parts. The second part includes the Dialysis Symptom Index (DSI) questionnaire to monitor disease specific burden from the perspective of patients (with a score ranging from 0-30, with a higher score defined as a higher disease burden). Scores before and after vaccination will be compared.
Change in behaviour towards measures against COVID-19 | two years
  Estimated by questionnaires, created by the studyteam in collaboration with the Dutch patient association. This questionnaire is focused on mental aspect of COVID-19 measures and whether certain measures, results or extra vaccinations influence behaviour of patients

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Stephan F Sanders, MD PhD, Study Director — University Medical Center Groningen; Marc H Hemmelder, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ahn C, Amer H, Anglicheau D, Ascher NL, Baan CC, Battsetset G, Bat-Ireedui B, Berney T, Betjes MGH, Bichu S, Birn H, Brennan D, Bromberg J, Caillard S, Cannon RM, Cantarovich M, Chan A, Chen ZS, Chapman JR, Cole EH, Cross N, Durand F, Egawa H, Emond JC, Farrero M, Friend PJ, Geissler EK, Ha J, Haberal MA, Henderson ML, Hesselink DA, Humar A, Jassem W, Jeong JC, Kaplan B, Kee T, Kim SJ, Kumar D, Legendre CM, Man K, Moulin B, Muller E, Munkhbat R, Od-Erdene L, Perrin P, Rela M, Tanabe K, Tedesco Silva H, Tinckam KT, Tullius SG, Wong G. Global Transplantation COVID Report March 2020. Transplantation. 2020 Oct;104(10):1974-1983. doi: 10.1097/TP.0000000000003258. No abstract available. PMID 32243281
- [Result] Baric RS. Emergence of a Highly Fit SARS-CoV-2 Variant. N Engl J Med. 2020 Dec 31;383(27):2684-2686. doi: 10.1056/NEJMcibr2032888. Epub 2020 Dec 16. No abstract available. PMID 33326716
- [Result] Robison SF, Mayhew RB, Cowan RD, Hawley RJ. Comparative study of deflection characteristics and fragility of 25-, 27-, and 30-gauge short dental needles. J Am Dent Assoc. 1984 Dec;109(6):920-4. doi: 10.14219/jada.archive.1984.0246. No abstract available. PMID 6595298
- [Result] Berends SE, Bloem K, de Vries A, Schaap T, Rispens T, Strik AS, Talwar R, Lowenberg M, D'Haens GR, Mathot RA. Monitoring of Adalimumab Concentrations at Home in Patients with Inflammatory Bowel Disease Using Dried Blood Samples. Ther Drug Monit. 2020 Apr;42(2):289-294. doi: 10.1097/FTD.0000000000000686. PMID 31464823
- [Result] Dearlove B, Lewitus E, Bai H, Li Y, Reeves DB, Joyce MG, Scott PT, Amare MF, Vasan S, Michael NL, Modjarrad K, Rolland M. A SARS-CoV-2 vaccine candidate would likely match all currently circulating variants. Proc Natl Acad Sci U S A. 2020 Sep 22;117(38):23652-23662. doi: 10.1073/pnas.2008281117. Epub 2020 Aug 31. PMID 32868447
- [Result] ERA-EDTA Council; ERACODA Working Group. Chronic kidney disease is a key risk factor for severe COVID-19: a call to action by the ERA-EDTA. Nephrol Dial Transplant. 2021 Jan 1;36(1):87-94. doi: 10.1093/ndt/gfaa314. PMID 33340043
- [Result] Gansevoort RT, Hilbrands LB. CKD is a key risk factor for COVID-19 mortality. Nat Rev Nephrol. 2020 Dec;16(12):705-706. doi: 10.1038/s41581-020-00349-4. PMID 32848205
- [Result] Gezondheidsraad. Strategieën voor COVID-19-vaccinatie. Den Haag: Gezondheidsraad, 2020; publicatienr. 2020/23
- [Result] Hilbrands LB, Duivenvoorden R, Vart P, Franssen CFM, Hemmelder MH, Jager KJ, Kieneker LM, Noordzij M, Pena MJ, Vries H, Arroyo D, Covic A, Crespo M, Goffin E, Islam M, Massy ZA, Montero N, Oliveira JP, Roca Munoz A, Sanchez JE, Sridharan S, Winzeler R, Gansevoort RT; ERACODA Collaborators. COVID-19-related mortality in kidney transplant and dialysis patients: results of the ERACODA collaboration. Nephrol Dial Transplant. 2020 Nov 1;35(11):1973-1983. doi: 10.1093/ndt/gfaa261. PMID 33151337
- [Result] Hodgson SH, Mansatta K, Mallett G, Harris V, Emary KRW, Pollard AJ. What defines an efficacious COVID-19 vaccine? A review of the challenges assessing the clinical efficacy of vaccines against SARS-CoV-2. Lancet Infect Dis. 2021 Feb;21(2):e26-e35. doi: 10.1016/S1473-3099(20)30773-8. Epub 2020 Oct 27. PMID 33125914
- [Result] Katerinis I, Hadaya K, Duquesnoy R, Ferrari-Lacraz S, Meier S, van Delden C, Martin PY, Siegrist CA, Villard J. De novo anti-HLA antibody after pandemic H1N1 and seasonal influenza immunization in kidney transplant recipients. Am J Transplant. 2011 Aug;11(8):1727-33. doi: 10.1111/j.1600-6143.2011.03604.x. Epub 2011 Jun 14. PMID 21672157
- [Result] Kotton CN. Immunization after kidney transplantation-what is necessary and what is safe? Nat Rev Nephrol. 2014 Oct;10(10):555-62. doi: 10.1038/nrneph.2014.122. Epub 2014 Jul 29. PMID 25072119
- [Result] Mahase E. Covid-19: Vaccine candidate may be more than 90% effective, interim results indicate. BMJ. 2020 Nov 9;371:m4347. doi: 10.1136/bmj.m4347. No abstract available. PMID 33168562
- [Result] Noordzij M, Duivenvoorden R, Pena MJ, de Vries H, Kieneker LM; collaborative ERACODA authors. ERACODA: the European database collecting clinical information of patients on kidney replacement therapy with COVID-19. Nephrol Dial Transplant. 2020 Dec 4;35(12):2023-2025. doi: 10.1093/ndt/gfaa179. No abstract available. PMID 32785669
- [Result] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Result] Reddy S, Chitturi C, Yee J. Vaccination in Chronic Kidney Disease. Adv Chronic Kidney Dis. 2019 Jan;26(1):72-78. doi: 10.1053/j.ackd.2018.10.002. PMID 30876620
- [Result] van der Willik EM, Meuleman Y, Prantl K, van Rijn G, Bos WJW, van Ittersum FJ, Bart HAJ, Hemmelder MH, Dekker FW. Patient-reported outcome measures: selection of a valid questionnaire for routine symptom assessment in patients with advanced chronic kidney disease - a four-phase mixed methods study. BMC Nephrol. 2019 Sep 2;20(1):344. doi: 10.1186/s12882-019-1521-9. PMID 31477039
- [Result] van Besouw NM, Yan L, de Kuiper R, Klepper M, Reijerkerk D, Dieterich M, Roelen DL, Claas FHJ, Clahsen-van Groningen MC, Hesselink DA, Baan CC. The Number of Donor-Specific IL-21 Producing Cells Before and After Transplantation Predicts Kidney Graft Rejection. Front Immunol. 2019 Apr 9;10:748. doi: 10.3389/fimmu.2019.00748. eCollection 2019. PMID 31024571
- [Result] Williamson EJ, Walker AJ, Bhaskaran K, Bacon S, Bates C, Morton CE, Curtis HJ, Mehrkar A, Evans D, Inglesby P, Cockburn J, McDonald HI, MacKenna B, Tomlinson L, Douglas IJ, Rentsch CT, Mathur R, Wong AYS, Grieve R, Harrison D, Forbes H, Schultze A, Croker R, Parry J, Hester F, Harper S, Perera R, Evans SJW, Smeeth L, Goldacre B. Factors associated with COVID-19-related death using OpenSAFELY. Nature. 2020 Aug;584(7821):430-436. doi: 10.1038/s41586-020-2521-4. Epub 2020 Jul 8. PMID 32640463
- [Derived] Vervoort JPM, Konijn WS, Jansen DEMC, Boersma C, de Zeeuw J, Ho-Dac-Pannekeet MM, Gansevoort RT, Messchendorp AL, Sanders JSF, de Wildt-Liesveld R. Patient engagement as a collaborative process in a large Dutch COVID-19 vaccination study (RECOVAC) - insight into the contribution of patient engagement and learnings for the future. Res Involv Engagem. 2024 Sep 13;10(1):96. doi: 10.1186/s40900-024-00622-x. PMID 39272117
- [Derived] Frolke SC, Bouwmans P, Messchendorp AL, Vervoort JPM, Abrahams AC, de Vries APJ, Nieuwkerk PT, Hemmelder MH, Gansevoort RT, Hilbrands LB, Reinders MEJ, Sanders JF, Bemelman FJ, Geerlings SE; RECOVAC Collaborators. Adherence to preventive measures after SARS-CoV-2 vaccination and after awareness of antibody response in kidney transplant recipients in the Netherlands: a nationwide questionnaire study. EClinicalMedicine. 2023 Jul 20;62:102103. doi: 10.1016/j.eclinm.2023.102103. eCollection 2023 Aug. PMID 37533418
- [Derived] Bouwmans P, Messchendorp AL, Sanders JS, Hilbrands L, Reinders MEJ, Vart P, Bemelman FJ, Abrahams AC, van den Dorpel MA, Ten Dam MA, de Vries APJ, Rispens T, Steenhuis M, Gansevoort RT, Hemmelder MH; RECOVAC Collaborators. Long-term efficacy and safety of SARS-CoV-2 vaccination in patients with chronic kidney disease, on dialysis or after kidney transplantation: a national prospective observational cohort study. BMC Nephrol. 2022 Feb 5;23(1):55. doi: 10.1186/s12882-022-02680-3. PMID 35123437